CLINICAL TRIAL: NCT04111172
Title: A Phase 2A, Dose-Finding Study of Ad5.F35-hGCC-PADRE Vaccine in Adults With Gastrointestinal Adenocarcinomas at Risk of Relapse Post Definitive Surgery and Standard Therapy
Brief Title: A Vaccine (Ad5.F35-hGCC-PADRE) for the Treatment of Gastrointestinal Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19P.785; JT 14133 (Other: JeffTrial Number)
Record Dates: First submitted 2019-09-20; First posted 2019-10-01 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Colorectal Adenocarcinoma; Gastric Adenocarcinoma; Clinical Stage II Gastric Cancer AJCC v8; Clinical Stage IIA Gastric Cancer AJCC v8; Clinical Stage IIB Esophageal Adenocarcinoma AJCC v8; Clinical Stage IIB Gastric Cancer AJCC v8; Clinical Stage III Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Gastric Cancer AJCC v8; Malignant Solid Neoplasm; Pathologic Stage II Gastric Cancer AJCC v8; Pathologic Stage IIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIB Gastric Cancer AJCC v8; Pathologic Stage III Esophageal Adenocarcinoma AJCC v8; Pathologic Stage III Gastric Cancer AJCC v8; Pathologic Stage IIIA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIA Gastric Cancer AJCC v8; Pathologic Stage IIIB Gastric Cancer AJCC v8; Pathologic Stage IIIC Gastric Cancer AJCC v8; Stage I Pancreatic Cancer AJCC v8; Stage IA Pancreatic Cancer AJCC v8; Stage IB Pancreatic Cancer AJCC v8; Stage II Pancreatic Cancer AJCC v8; Stage IIA Pancreatic Cancer AJCC v8; Stage IIB Pancreatic Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Malignant Digestive System Neoplasm; Small Intestinal Adenocarcinoma; Stage III Small Intestinal Adenocarcinoma AJCC v8; Stage IIIA Small Intestinal Adenocarcinoma AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (low dose) (Experimental): Patients receive low dose Ad5.F35-hGCC-PADRE vaccine IM on day 1 of weeks 1, 5, and 9 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Adenovirus 5/F35-Human Guanylyl Cyclase C-PADRE
- Arm B (medium dose) (Experimental): Patients receive medium dose Ad5.F35-hGCC-PADRE vaccine IM on day 1 of weeks 1, 5, and 9 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Adenovirus 5/F35-Human Guanylyl Cyclase C-PADRE
- Arm C (high dose) (Experimental): Patients receive high dose Ad5.F35-hGCC-PADRE vaccine IM on day 1 of weeks 1, 5, and 9 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Adenovirus 5/F35-Human Guanylyl Cyclase C-PADRE

INTERVENTIONS:
Biological: Adenovirus 5/F35-Human Guanylyl Cyclase C-PADRE — Given as intramuscular injection
  Other Names: Ad5.F35-hGCC-PADRE; Ad5/F35-hGCC-PADRE; Adenovirus 5/F35-HGCC-PADRE

SUMMARY:
This phase IIA trial investigates the side effects of Ad5.F35-hGCC-PADRE vaccine and to see how well it works in treating patients with gastrointestinal adenocarcinoma. Ad5.F35-hGCC-PADRE vaccine may help to train the patient's own immune system to identify and kill tumor cells and prevent it from coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of sequential adenovirus 5/F35-human guanylyl cyclase C-PADRE (Ad5.F35-hGCC-PADRE), delivered intramuscularly three times at three dose levels in subjects with high-risk colorectal, pancreatic, gastric, or esophageal adenocarcinomas with no evidence of disease (NED) after surgery and standard therapy.

II. Evaluate the cellular (T-cell) responses to Ad5.F35-hGCC-PADRE at three different dose levels (10^11, 10^12, and 5 x 10^12 vp) administered intramuscularly three times, four weeks apart in subjects with high-risk colorectal, pancreatic, gastric, or esophageal cancer with NED after surgery and standard therapy.

EXPLORATORY OBJECTIVES:

I. Evaluate the humoral immunologic response to guanylyl cyclase C (GCC), defined as an incremental or sustained antibody (pan-Ig) response, measured at weeks 5, 9, and 13 following the first vaccination (week 1).

II. Evaluate the relationship between immunological responses to GCC and 1) neutralizing antibodies to Ad5 and Ad5.F35 and 2) GCC protein expression in tumors to assess immune tolerance.

III. Evaluate disease free survival (DFS) and overall survival (OS), where feasible.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM A: Patients receive low dose Ad5.F35-hGCC-PADRE vaccine intramuscularly (IM) on day 1 of weeks 1, 5, and 9 in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive medium dose Ad5.F35-hGCC-PADRE vaccine IM on day 1 of weeks 1, 5, and 9 in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive high dose Ad5.F35-hGCC-PADRE vaccine IM on day 1 of weeks 1, 5, and 9 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 28 days, and then every 3 months for at least 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Subjects with tumors specified below, who are at high risk of relapse, have been treated with curative intent, and have no evidence of disease (NED) following front-line therapy with surgery, radiation therapy, and/or chemotherapy. NED includes, where applicable, surgical (macroscopic tumor margin, at the time of surgery), and radiological evidence of disease. Residual lesions identified by microscopic/frozen margins and biochemical markers are permitted. Therapy must have been completed no fewer than four weeks, and no later than 25 weeks, before the first dose of Ad5.F35-hGCC-PADRE
* For tumor-specific criteria, please refer to the information below:

  * Pancreatic ductal adenocarcinoma

  ** Stage I, II, III
  * Neuroendocrine tumors of the pancreas are not permitted

    * Colorectal adenocarcinoma
    * Stage III; stage IV following metastasectomy

      * Gastric adenocarcinoma
    * Stage IIA, IIB, III
  * Gastrointestinal stromal tumors of the stomach are not permitted

    * Esophageal adenocarcinoma

    ** Stage IIB, III
  * Esophageal squamous cell carcinomas are not permitted
* Have an anticipated life expectancy of greater than 12 weeks
* Absolute neutrophil count (ANC) >= 1000 cells/mL
* Platelets >= 75,000 /mL
* Hemoglobin >= 9.0 g/dL
* Serum creatinine < 2.0 mg/dL
* For other blood and urine tests including blood chemistry, hepatic and renal functions, test results should not be worse than grade 1 levels of abnormalities defined by Common Terminology Criteria for Adverse Events (CTCAE), National Cancer Institute (NCI) version 5 issued by the United States (US) Department of Health and Human Services
* For women and men of childbearing potential, a medically acceptable method of highly effective contraception (oral hormonal contraceptive, condom plus spermicide, or hormonal implants) or abstinence must be used throughout the study period and for 28 days after their final vaccine administration (a barrier method of contraception must be employed by all subjects [male and female], regardless of other methods unless abstinent). A negative serum or urine pregnancy test is required as part of screening. Women of childbearing potential is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/ml
* Be willing to comply with all the study procedures
* All subjects must be able to comprehend and sign a written informed consent document

Exclusion Criteria:

* Have a known history or evidence of residual disease after definitive surgery
* Have a known metastasis in the brain or central nervous system
* Prior receipt of immunotherapy or experimental medications after completion of standard adjuvant therapy
* Have a history of splenectomy
* Have a history of distal pancreatectomy
* Concurrent use of systemic steroids or immunosuppressive drugs (use of topical or inhaled steroids will be allowed)
* Have any immunodeficiency disease or immunocompromised state (e.g., use of immunosuppressive agents, chemotherapy or radiation therapy within four weeks of study treatment)
* Have active autoimmune disease or history of autoimmune disease or a transplant recipient requiring systemic steroids or other immunosuppressive treatment
* Have received a diagnosis of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C (subjects who are hepatitis C positive may be enrolled if they are confirmed with negative viral load at screening)
* Other malignancy within last 5 years except curatively treated non-melanomatous skin cancer and curatively treated carcinoma in situ of the uterine cervix, or early-stage (stage A or B1) prostate cancer
* Have a history of inflammatory bowel disease
* Have a history of serious reaction to adenovirus
* Have an intercurrent illness that is either life-threatening or of clinical importance such that it might limit study compliance (such illnesses include, but are not limited to, ongoing or active infection, metabolic or neurologic disease, peripheral vascular disease, or psychiatric illness)
* Have insufficient peripheral venous access to permit completion of the study phlebotomy regimen
* Consumes greater than three glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce]) per day and cannot refrain from alcohol for the duration of the trial
* Has a history of use of illicit drugs (e.g., opioids, cocaine, amphetamines, hallucinogens, etc.) that could potentially interfere with adherence to study procedures or requirements
* Be a woman who is pregnant or breastfeeding
* Have an unhealed surgical wound
* Have had major surgery or significant traumatic injury occurring within 28 days before treatment or anticipated surgery or procedure requiring general anesthesia during the study participation (including four weeks after last dose of vaccine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 13 weeks
  AEs classified by System Organ Class, preferred term, severity, and relationship to study treatment, and graded in accordance with the document entitled "Common Terminology Criteria for Adverse Events" (CTCAE), National Cancer Institute version 5 issued by the United States Department of Health and Human Services. Injection-site reactions including, but not necessarily limited to, local skin erythema, induration, pain and tenderness at administration site. Clinically-significant changes in safety laboratory tests. The percentage of subjects with AEs and DLTs will be summarized along with corresponding 95% confidence intervals for each treatment arm and overall.
Antigen-specific T-cell response to guanylyl cyclase C (GCC) | 13 weeks
  Will be measured by enzyme-linked immunosorbent spot (ELISpot) assay. the immune parameters will be summarized via percentages of responders and mean/median values, along with corresponding 95% confidence intervals, by treatment arm and measurement time. Antibody and T-cell data will be summarized by positive response rates (each subject recorded as yes/no) and exact 2-sided 95% confidence intervals. For this study, a statistically significant increase in GCC-specific T-cell response at Weeks 5, 9, or 13 compared with baseline will be considered a response at that time. Significance of the change from baseline will be assessed using the modified distribution-free resampling (DFR) method. Will estimate response rates across disease types.

CONTACTS AND LOCATIONS:
Overall Officials: Babar Bashir, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No